CLINICAL TRIAL: NCT00132886
Title: Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Single Oral Tolvaptan Tablets on Hemodynamic Parameters in Subjects With Heart Failure
Brief Title: Heart Pressure Assessment Study With Tolvaptan to Treat Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-04-247
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

INTERVENTIONS:
Drug: tolvaptan

SUMMARY:
This study will look at how a single dose of study medication (tolvaptan) versus an inactive sugar pill (placebo) effect pressures in the heart in patients with congestive heart failure. Higher than normal pressures can be related to symptoms of heart failure (shortness of breath, fatigue, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Class III or IV heart failure for at least 3 months
* Left ventricular ejection fraction less than or equal to 40%
* Currently being treated for heart failure with standard therapies for at least one month

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Inability to take oral medications
* Uncontrolled hypertension, bradyarrhythmias or tachyarrhythmias
* Hypertrophic obstructive cardiomyopathy
* Severe obstructive pulmonary disease
* Significant renal impairment
* Significant uncorrected valvular or congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in heart pressures (PCWP) at 3 to 8 hours post-dose

SECONDARY OUTCOMES:
Change in heart function measurements (CI, SVR, PVR, RAP) at 3 to 8 hours post-dose
Change in urine output and free water clearance
Change from baseline in urine osmolality
Cmax, tmax, and AUC 12h of tolvaptan in plasma
Adverse events, vital signs and clinical labs

CONTACTS AND LOCATIONS:
Overall Officials: James Udelson, MD, Study Chair — Cardiovascular Clinical Studies and Tufts/New England Medical Center
Locations (31):
- United States (26):
  - Oracle Research, A Div of the Heart Center, Huntsville, Alabama
  - Merced Heart Associates, Merced, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Cardiovascular Center at Shands Jacksonville, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - ACRI, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Robert Rush University Medical Center, Chicago, Illinois
  - Loyola University of Chicago, Maywood, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Cardiologist Institute, Slidell, Louisiana
  - Medical Research Institute Louisiana Heart Hospital, Slidell, Louisiana
  - Primary Cardiology Associates, Ayer, Massachusetts
  - U-MASS Memorial Medical Center, Worchester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Heart Consultants, PC, Omaha, Nebraska
  - University of Medicine and Dentistry, Newark, New Jersey
  - UNC Heart Failure Program, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland VA Medical Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Guthrie Foundation, Syre, Pennsylvania
  - Texas Heart Institute, Houston, Texas
  - Southeast Texas Clinical Research, Orange, Texas
- Romania (5):
  - Spitalul Clinic Urgenta, Bucharest
  - Institutul de Boli Cardiovasculare, Bucharest
  - Institutul de Boli Cardiovasculare"Prof. Dr. C.C. Illiescu", Bucharest
  - Institutul Inimii, Judetul Cluj
  - Institutul de Boli Cardiovasculare si Transplant, Judetul Mures

REFERENCES:
- [Derived] Hiukka A, Westerbacka J, Leinonen ES, Watanabe H, Wiklund O, Hulten LM, Salonen JT, Tuomainen TP, Yki-Jarvinen H, Keech AC, Taskinen MR. Long-term effects of fenofibrate on carotid intima-media thickness and augmentation index in subjects with type 2 diabetes mellitus. J Am Coll Cardiol. 2008 Dec 16;52(25):2190-7. doi: 10.1016/j.jacc.2008.09.049. PMID 19095138
- [Derived] Udelson JE, Orlandi C, Ouyang J, Krasa H, Zimmer CA, Frivold G, Haught WH, Meymandi S, Macarie C, Raef D, Wedge P, Konstam MA, Gheorghiade M. Acute hemodynamic effects of tolvaptan, a vasopressin V2 receptor blocker, in patients with symptomatic heart failure and systolic dysfunction: an international, multicenter, randomized, placebo-controlled trial. J Am Coll Cardiol. 2008 Nov 4;52(19):1540-5. doi: 10.1016/j.jacc.2008.08.013. PMID 19007589